CLINICAL TRIAL: NCT03090841
Title: Biomarkers of Fetal Infection and Disease Following Maternal HCMV Infection
Brief Title: Biomarkers of Cytomegalovirus Fetal Infection and Disease
Acronym: BIO-CCMV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 14024
Record Dates: First submitted 2017-01-03; First posted 2017-03-27 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Cytomegalovirus Congenital
Keywords: Cytomegalovirus Congenital; Non-invasive diagnosis; Omics; Biomarkers
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Amniotic fluid (2ml)
  * Fetal blood (2 ml)
  * Maternal blood (5 ml)
  * Cord blood (50 ml)
  * Neonatal blood (2 ml)
  * Neonatal urine (2 ml
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CMV cases: bio-specimen collected for pregnant women with CMV infection
  Interventions: Biological: Bio-specimen collected
- Control cases: bio-specimen collected for pregnant women carrying a fetus with aneuploidy-dysgonosomy
  Interventions: Biological: Bio-specimen collected

INTERVENTIONS:
Biological: Bio-specimen collected

SUMMARY:
The purposes of this study are to determine 1) if the diagnosis of CMV fetal infection could be done directly in the maternal blood instead of requesting an amniocentesis and 2) if innovative technologies such as proteomic, transcriptomic, methylomic and lipidomic applied in fetal samples could allow the discovery of new biomarkers of fetal infection.

DETAILED DESCRIPTION:
Human cytomegalovirus (HCMV) is the most common cause of congenital infection worldwide. The diagnosis of CMV fetal infection relies on the detection of viral DNA in amniotic fluid by polymerase chain reaction after amniocentesis. Non-invasive diagnosis of fetal infection directly in maternal blood is not available. Symptoms develop in about 10% of HCMV-infected fetuses. Despite important advance in medical imaging, establishing the prognosis of an infected fetus remains challenging. Thrombocytopenia, blood HCMV DNA, anti-HCMV immunoglobulin M and β2-microglobulin are recognized biomarkers of symptomatic fetal infections. However, the predictive value of these individual markers is not. Omics technologies could help to establish multimarker signatures of symptomatic infections.

The objective of the study is to:

* validate fetal blood HCMV DNA, anti-HCMV immunoglobulin M , β2-microglobulin and platelet count as biomarkers of fetal disease;
* identify new biomarkers of severe fetal disease using transcriptomic, methylomic and lipidomic analyses of fetal blood and of amniotic fluid.
* validate a non-invasive CMV fetal infection diagnosis tool based on deep-sequencing of targeted CMV genes in maternal blood

ELIGIBILITY:
Inclusion Criteria:

CMV cases:

* Informed consent obtained from the mother;
* Pregnant women either with a history of primary CMV infection in pregnancy or carrying a fetus with ultrasound features compatible with CMV infection and willing to have amniocentesis for fetal diagnosis of CMV infection

Control cases :

- Pregnant women carrying a fetus with aneuploidy-dysgonosomy

Exclusion Criteria:

CMV cases:

* Fetuses older than the 26 weeks of gestation at the time of diagnosis of HCMV infection or impossibility to collect foetal samples by the end of the 26th week of gestation
* Mother unable to understand the protocol
* Absence of informed consent
* Any clinical rationale not to perform cordocentesis
* Mother <18 years age
* Administration of immunoglobulins or anti-viral therapy to the mother before the collection of fetal samples or before the diagnosis of symptomatic fetal infection
* Administration of anti-HCMV drugs to the foetus before the collection of fetal samples or before the diagnosis of symptomatic fetal infection
* Administration of immunosuppressive drugs to the mother during pregnancy
* Maternal auto immune disorders
* Multiple pregnancies.

Control cases :

* Mother unable to understand the protocol
* Absence of informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 320 pregnant women with CMV primary infection or carrying a fetus with compatible ultrasound features to obtained 65 infected fetuses and 15 fetuses diagnosed with severely symptomatic infection
  * 200 controls pregnant women carrying a fetus with aneuploidy-dysgonosomy
Sampling Method: Non-Probability Sample
Enrollment: 265 (Estimated)
Dates: Start 2016-12; Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values in fetal blood | At 23 weeks gestation +/- 3 weeks
  Fetal platelet in mm3/ml, β2 microglobulinein mg/L, proteins concentration in mg/L , Metabolites concentration in mmoles/l , Lipids concentration in mmoles/l , RNA messagers concentration in µg/ml profil

SECONDARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values in amniotic fluid | At 23 weeks gestation +/- 3 weeks
  CMV DNA quantification in UI/mL , protein concentration in mg/L, Metabolites concentration in mmoles/l , Lipids concentration in mmoles/l, RNAm concentration in µg/ml profil ,
Non invasive diagnosis of fetal CMV infection in maternal blood in UI/mL. | At 23 weeks gestation +/- 5 weeks
  CMV fetal DNA measurement in maternal blood

CONTACTS AND LOCATIONS:
Overall Officials: Yves VILLE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants-Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benoist G, Salomon LJ, Jacquemard F, Daffos F, Ville Y. The prognostic value of ultrasound abnormalities and biological parameters in blood of fetuses infected with cytomegalovirus. BJOG. 2008 Jun;115(7):823-9. doi: 10.1111/j.1471-0528.2008.01714.x. PMID 18485159
- [Background] Fabbri E, Revello MG, Furione M, Zavattoni M, Lilleri D, Tassis B, Quarenghi A, Rustico M, Nicolini U, Ferrazzi E, Gerna G. Prognostic markers of symptomatic congenital human cytomegalovirus infection in fetal blood. BJOG. 2011 Mar;118(4):448-56. doi: 10.1111/j.1471-0528.2010.02822.x. Epub 2010 Dec 24. PMID 21199291
- [Background] Desveaux C, Klein J, Leruez-Ville M, Ramirez-Torres A, Lacroix C, Breuil B, Froment C, Bascands JL, Schanstra JP, Ville Y. Identification of Symptomatic Fetuses Infected with Cytomegalovirus Using Amniotic Fluid Peptide Biomarkers. PLoS Pathog. 2016 Jan 25;12(1):e1005395. doi: 10.1371/journal.ppat.1005395. eCollection 2016 Jan. PMID 26808779
- [Derived] Bourgon N, Fitzgerald W, Aschard H, Magny JF, Guilleminot T, Stirnemann J, Romero R, Ville Y, Margolis L, Leruez-Ville M. Cytokine Profiling of Amniotic Fluid from Congenital Cytomegalovirus Infection. Viruses. 2022 Sep 28;14(10):2145. doi: 10.3390/v14102145. PMID 36298700